CLINICAL TRIAL: NCT02671617
Title: A Randomised Control Trial to Assess Efficacy of Preoperative High Intensity Interval Training in Elderly Patients Scheduled for Oncological Abdominal Surgery
Brief Title: Preoperative HIIT in Elderly Cancer Patients
Acronym: eHIITCa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: eHIITCa
Record Dates: First submitted 2016-01-18; First posted 2016-02-02 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Cancer
Keywords: Abdominal Cavity; Aged
MeSH Terms: conditions — Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control: This group of patients will receive 'current best practice' as per UK NHS recommendations for their specific cancer management prior to surgery.
- High intensity interval training (Experimental): Exercise: Participants in this group will attend 3-4 times per week to complete HIIT training during the period from diagnosis to surgery.
  High intensity interval training (HIIT)
  Interventions: Other: High intensity interval training (HIIT)

INTERVENTIONS:
Other: High intensity interval training (HIIT) — Preoperative HIIT protocol.
  Arms: High intensity interval training

SUMMARY:
This randomized control trial will determine the effect of short term high intensity interval training (HIIT) on physical fitness, in an elderly patient group with active cancer, prior to surgical resection.

Half of the recruited patients will act as a control group and the other half will undergo a HIIT protocol.

DETAILED DESCRIPTION:
High intensity interval training (HIIT) has been shown to achieve similar and in some studies better improvements in aerobic fitness versus more traditional endurance based exercise over the same time period. HIIT has also been shown to produce these improvements over a shorter timescale than other methods, in the region of 2-6 weeks. One widely reported barrier to exercise is time availability, HIIT training may be a favorable option to increase fitness as the total time spent exercising is significantly less than other methods. HIIT induces improvements in cardiovascular parameters in healthy elderly subjects, investigators aim to investigate whether these improvements can be matched in patients with cancer and further elucidate the mechanisms behind improvements seen with this type of training.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years (no upper age limit).
* Histologically proven, radiologically or direct visualisation leading to high clinical suspicion of cancer.
* Sufficient mobility to be able to exercise on a static exercise bike.
* Ability to give informed consent.
* Ability to travel to RDH to complete the HIIT sessions (may also rely upon dependents/relatives to provide transport).

Exclusion Criteria:

* Adjuvant systemic chemotherapy / radiotherapy treatment for this cancer. Participants with a significant past medical history of:
* Myocardial infarction (within last 6 months)
* Unstable Angina
* Heart failure (NYHA class III/IV)
* Uncontrolled Hypertension (BP>160/100)
* Previous stroke/TIA
* Severe respiratory disease inc. known pulmonary hypertension(>25 mmHg), Forced Expiratory Volume in 1 second <1.5l.
* Brittle asthma / exercise induced asthma
* Known cerebral aneurysm.
* Inclusion in a recent (within 3 months) study which included any form of exercise, taking a drug or ionising radiation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
VO2AT (VO2 at anaerobic threshold) | Baseline and 4 weeks
  Change in anaerobic threshold seen during maximal exercise test (pre and post intervention).

SECONDARY OUTCOMES:
VO2peak | Baseline and 4 weeks
  Change in peak volume of oxygen consumption during maximal exercise test (pre and post intervention).
Subjective acceptability of HIIT preoperatively (via questionnaire) | After 4 weeks of HIIT.
  Assessment of whether our HIIT protocol is acceptable to patients in this age group.
Muscle protein synthesis rate changes with HIIT. | Baseline and 4 weeks.
  Assessment of the effect HIIT has on rate of muscle protein synthesis in this group.

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, MBChB FRCA PhD, Principal Investigator — Nottingham University
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be made available.